CLINICAL TRIAL: NCT06789991
Title: Electromyographic Activity of Posterior Oblique Sling Muscles in Patients With Shoulder Impingement Syndrome
Acronym: EMG
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nada mohamed ahmed emara, principle investigator, Cairo University
Other Study IDs: P.T.REC/012/005452; P.T.REC/012/005452 (Other: ethical committee faculty of physical therapy CU)
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A (control group): controls
  Interventions: Device: electromyography
- Group B (experimental group): cases
  Interventions: Device: electromyography

INTERVENTIONS:
Device: electromyography — electromyographic activity of posterior oblique sling muscles will be measured

SUMMARY:
this study aims to assess the gluteus maximus muscle electromyographic activity and the latissimus dorsi muscle electromyographic activity in patients with shoulder impingement syndrome , to improve the assessment procedure and the rehabilitation program for treating patients with shoulder impingement syndrome more effectively. .

DETAILED DESCRIPTION:
background: Shoulder pain is the third most common musculoskeletal complaint that can lead to disability that interfere with work, hobbies, social, and sporting activities and may also be associated with psychological distress and reduced quality of life .Shoulder impingement syndrome Symptoms is the most common cause of shoulder pain.

Normal shoulder movement is achieved through a stable lumbopelvic-hip complex and scapula. Thus, the pelvis must provide a stable platform for the scapula and the scapula provide a stable platform for the shoulder. The existing evidence supports myofascial biomechanical connection between lumbopelvic region and contralateral glenohumeral joint .So Considering the LP region and related myofascial force transmission as contributing factors for shoulder pathogenesis can explain the reasoning on why some of the patients with shoulder pain may progress to develop chronic shoulder pain.

purpose: this study aims to assess the gluteus maximus muscle electromyographic activity and the latissimus dorsi muscle electromyographic activity in patients with shoulder impingement syndrome , to improve the assessment procedure and the rehabilitation program for treating patients with shoulder impingement syndrome more effectively.

methods: This study is a cross sectional comparative study will be conducted at the out-patient physical therapy clinic, Pharos University in Alexandria, Egypt. 30 patients with unilateral shoulder impingement and 30 healthy controls without shoulder impingement , with age range between 25 and 40 years will be included in the study. All patients will be referred by an orthopedic surgeon.

results: data analysis with one-way ANOVA will be used to compare between subjects characteristics of the two groups and un-paired t-test will be used to compare measured variables between groups.

keywords: shoulder impingement syndrome, posterior oblique sling , electromyography , latissimus dorsi , gluteus maximus

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients with shoulder impingement syndrome.
2. patients complain from unilateral shoulder pain with chronic conditions of SIS ≥ 3 months.
3. Patient age from 25 to 40 years.
4. Patients with Positive impingement tests.
5. Patients with painful arc of movement (60°- 120°)

Exclusion Criteria:

1. Patients with Numbness or tingling of upper extremity.
2. Patients with Shoulder fracture or previous shoulder surgery, and Acromioclavicular or shoulder dislocation.
3. Patients with Any traumatic injury to the lower limb in the previous 6 months.
4. Any spine surgery within the last 2 years.
5. Patients with history of lower back pain in past 12 months .
6. Patients with history of lower extremity dysfunctions in the past 12 months .
7. Participants who had taken any drugs (e.g. statins and spasmed), which have effects on the skeletal muscles.
8. Open wounds, rashes, psoriasis, skin irritations, or skin conditions of any kind in the region of electrode placement
9. Participants with a Body Mass Index (BMI) ≥ 30

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients will be referred by an orthopedic surgeon who will diagnose SIS based on clinical and radiological examination.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
• electromyographic activity of posterior oblique sling muscles (gluteus maximus and latissimus dorsi) | through study completion, an average of 4 months
  EMG has been widely used for many decades, its use is proven and widely accepted by clinicians and the scientific community and it is considered the gold standard method for the measurement of muscle activity.

SECONDARY OUTCOMES:
shoulder active range of motion | through study completion, an average of 4 months
  Universal goniometry is frequently used by physical therapists to assess ROM due to its ease of use, portability, noninvasive nature, and low cost.
shoulder function and disability level | through study completion, an average of 4 months
  The Arabic Q-DASH questionnaire has demonstrated good reliability, validity, and responsiveness when used for patients with upper extremity disorders.
shoulder pain | through study completion, an average of 4 months
  The ordinal 11-point NPRS (0-no pain, 10-most intense pain) has good test-retest reliability (r=.79-.96) in individuals with chronic pain and musculoskeletal pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir S Rizk, PhD, Study Chair — Cairo University; Aya A Khalil, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No